CLINICAL TRIAL: NCT02227030
Title: Tolerability and Pharmacokinetics of Single Oral Administration of 10, 20, 50, 100, 200 and 300 mg BIIB 722 CL (Calculated as Free Base) as Drinking Solution and of 200, 450, 600 and 750 mg BIIB 722 CL as Filmcoated Tablet in Healthy Subjects. An Open Study With Rising Doses, Partly Uncontrolled Intra-individual Comparison, Placebo Randomised Double Blind at Each Dose Level.
Brief Title: Tolerability and Pharmacokinetics of BIIB 722 CL Drinking Solution and of BIIB 722 CL Filmcoated Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1180.1
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Solutions; Tablets

ARMS (4):
- BIIB 722 CL single rising dose (Experimental)
  Interventions: Drug: BIIB 722 CL solution
- BIIB 722 CL cross over (Experimental)
  Interventions: Drug: BIIB 722 CL solution; Drug: BIIB 722 CL tablet
- Placebo solution (Placebo Comparator)
  Interventions: Drug: Placebo solution
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: BIIB 722 CL solution
  Arms: BIIB 722 CL cross over; BIIB 722 CL single rising dose
Drug: BIIB 722 CL tablet
  Arms: BIIB 722 CL cross over
Drug: Placebo solution
  Arms: Placebo solution
Drug: Placebo tablet
  Arms: Placebo tablet

SUMMARY:
Safety and pharmacokinetics after oral single rising doses of BIIB 722 CL

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* 18 to 55 years of age
* Broca index >= -20% and <= +20%
* Written informed consent according to Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* History or current gastrointestinal hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs, which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2000-04; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma (AUC) | up to 96 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax) | up to 96 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 96 hours after drug administration
Total mean residence time of the analyte in the body (MRTtot) | up to 96 hours after drug administration
Total clearance of the analyte in plasma (CLtot/f) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 96 hours after drug administration
Number of subjects with clinically significant findings in vital functions | up to 96 hours after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 96 hours after drug administration
Thrombocytic Na-H exchange (NHE-1) inhibition by AUC of pH recovery | up to 24 hours after drug administration